CLINICAL TRIAL: NCT06252194
Title: Comparative Study of Metformin Versus Doxycycline in Treatment of Moderate to Severe Adult Acne Vulgaris Patients: Multicentre, Randomized, Double-blind Trial.
Brief Title: Comparative Study of Metformin Versus Doxycycline in Moderate to Severe Adult Acne Vulgaris Patients.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Marnush, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSMMU/2022/11379
Record Dates: First submitted 2024-01-30; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Metformin; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Metformin 500 mg twice daily along with topical retinoids for 12 weeks
  Interventions: Drug: Metformin and doxycycline
- Group B (Active Comparator): Doxycycline 100 mg twice daily along with topical retinoids for 12 weeks
  Interventions: Drug: Metformin and doxycycline

INTERVENTIONS:
Drug: Metformin and doxycycline — Metformin 500 mg tablet twice daily

SUMMARY:
The goal of this clinical trial is to compare the effect of doxycycline and metformin in treatment of acne vulgaris patients. The main question is aimed to answer is whether metformin is more effective than doxycycline in treatment of acne vulgaris patient or not.

Patients will be asked to take doxycycline along with tropical treatment in one group and metformin along with tropical treatment in another group.

Researcher will compare the clinical improvement in two groups.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed moderate and severe AV patients diagnosed by a dermatologist

-

Exclusion Criteria:

* Patients receiving topical retinoids within last two months
* Pregnancy and lactation
* History of corticosteroids intake
* Suffering from malignancy or any cosmetic induced acne

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Global Acne Grading System (GAGS) Score | 12 weeks
  Acne Vulgaris Severity assesment by GAGS score

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No